CLINICAL TRIAL: NCT05556915
Title: Intérêt De L'échoguidage Dans Les Ponctions De Fistule Artério-veineuse En Hémodialyse Pédiatrique
Brief Title: Benefit of Ultrasound Guidance in Arteriovenous Fistula (AVF) Cannulation in Pediatric Hemodialysis
Acronym: PafusGuC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL21_0526
Record Dates: First submitted 2022-09-13; First posted 2022-09-27 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Arteriovenous Fistula Cannulation
Keywords: Arteriovenous fistula AVF; Pediatric hemodialysis; Cannulation

STUDY DESIGN:
Intervention Model Description: Open label, randomized clinical study comparing two AVF cannulation methodes (conventional vs ultrasound-guided method) in pediatric patients with end-stage renal disease undergoing hemodialysis therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-guided AVF cannulation method (Experimental): The AVF cannulation is carried out using ultrasoud guidance
  Interventions: Other: Ultrasound-guided AVF cannulation method
- Conventional AVF cannulation method (Other): The AVF cannulation is carried out by palpation
  Interventions: Other: Conventional AVF cannulation method

INTERVENTIONS:
Other: Ultrasound-guided AVF cannulation method — For ultrasound-guided cannulation, the same ultrasound device will be used for all patients (TE5-POC ultrasound MINDRAY® system). The ultrasound device will identify the AVF aspect , the location including the depth (distance from the skin surface) , the vessel diameter and guide the cannulation in real-time. The device will be disinfected between uses and covered with a transparent adhesive film to avoid any direct contact with the patient. Sterile gel will be used for the cannulation.
  Arms: Ultrasound-guided AVF cannulation method
Other: Conventional AVF cannulation method — The AVF cannulation is carried out by palpation. This technique consists of manually evaluating the position, direction and depth of the fistula in order to determine the puncture site where the 2-dialysis catheters will be inserted. After local asepsis, the AVF is therefore needled at 2 points 5 cm apart.
  Arms: Conventional AVF cannulation method

SUMMARY:
The arteriovenous fistula (AVF) is the reference hemodialysis vascular access for both adult and pediatric patients. The cannulation quality is decisive for the quality of the dialysis. Difficult AVF cannulations are more frequent in pediatrics than in adults. Recent studies in adults have shown that ultrasound-guided AVF cannulation improves the cannulation quality and therefore the quality of dialysis. This study aims to prove that ultrasound-guided AVF cannulation in children will improve the quality of dialysis overall.

DETAILED DESCRIPTION:
The European and American recommandations emphasize that the arteriovenous fistula (AVF) is the first choice vascular access in hemodialysis for both adult and pediatric patients. Indeed, infections and thrombotic complications are lower with an AVF than with a central venous catheter. In addition, the efficiency of dialysis is better in patients with AVF in both pediatric and adult patients.

The pediatric population has its own characteristics. On the one hand, the size of the vessels, in particular in patients weighing less than 20 kilos, complicates the creation of the AVF. On the other hand, the time for AVF maturation in children (corresponding to the time required between the creation of the AVF and its use) is much higher than that of the adult population. These specific anatomical characteristics partly explain the more frequent AVF cannulation difficulties in pediatric patients.

Inadequate dialysis is considered to be a session in which the therapy goals were not achieved. This rate of inadequate dialysis is estimated at 8-10% in children due to vascular access problem, whereas this rate is only 1 to 5% in adults. There is also an increase in side effects related to these pediatric AVF cannulation difficulties (trauma, hematoma, edema following diffusion, etc.) responsible for inadequate dialysis and, in the long term, AVF dysfunction (stenosis, thrombosis).

The preservation of the vascular access by means of new cannulation techniques aimed at limiting trauma is therefore a primary objective in pediatric hemodialysis. The introduction of new cannulation methods as well as the training of nurses/childcare workers in the various puncture techniques would thus make it possible to improve the quality of dialysis sessions, the lifespan of AVFs, to increase the number of puncture sites and reduce the number of punctures per session and the occurrence of complications.

Recently, the ultrasound-guided AVF cannulation technique has shown promising results in adults with regard to the prevention of vascular access complications, the feeling of pain and the obtaining of adequate dialysis.

A recent review points to the need to confirm the benefit of ultrasound-guided cannulation through randomized studies, the current data being promising but needing to be confirmed. To date, no data concerning the benefit of ultrasound-guided cannulation in pediatrics is available in the literature. Our project will therefore be the first research to compare 2 AVF cannulation methods in pediatric hemodialysis. The hypothesis adopted is that the AVF cannulation using ultrasound guidance in children undergoing dialysis will allow an overall improvement of dialysis quality, a reduction of complication occurrence and an improvement of patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients ˂ 18 years of age at enrollment
* Patients with end-stage renal disease undergoing hemodialysis therapy
* Patients carrying an arteriovenous fistula created more than 6 weeks before enrollment
* Prior agreement of the patient and their legal representative by signing the parent's informed consent form
* Patients affiliated to social security system

Exclusion Criteria:

* Non-matured arteriovenous fistula according to the referring pediatrician
* Patients undergoing dialysis at least partly through a central venous catheter
* Estimated duration of dialysis less than 1 month in the investigation center
* Participation in other intervention research

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2022-12-03 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Compare the rate of inadequate dialysis after ultrasound-guided AVF cannulation vs. conventional cannulation in pediatric patients (<18 years) with end-stage renal disease undergoing hemodialysis therapy. | 12 months
  Inadequate dialysis is defined by the presence of one of the following parameters:
  * Blood flow rate (BFR expressed in ml/min corresponding to the volume of blood in milliliters that flows per minute) less than 80% of adequate blood flow corresponding to a flow ≥ 7 ml per kilograms of weight with a maximum of 300 ml/min
  * Requirement of single-needle dialysis after 3 cannulation failures
  * Early discontinuation of hemodialysis
  * Loss of dialysis circuit during the session
  * Out of range arterial or venous pressure during dialysis requiring a drop in blood flow rate
  * Purification coefficient defined by Kt/V <1.2: K represents the dialyzer clearance of urea (expressed in milliliters/ min and corresponds to the volume of blood in ml cleared of urea per minute ) // t (in minutes) represents the dialysis time duration // V (in milliliters) represents the volume of distribution of urea, and equals the patient's total body water

SECONDARY OUTCOMES:
Number of cannulations required for the insertion of the 2 dialysis catheters | During procedure
  Compare the number of cannulations required for the insertion of the 2 dialysis catheters in conventional method vs ultrasound-guided method
The time required for the insertion of the 2 catheters | During procedure
  Compare the time required for the insertion of the 2 catheters in conventional method vs ultrasound-guided method
The occurrence of cannulation complications | During procedure
  Compare the occurrence of cannulation complications (hematoma, diffusion, aneurysm, etc.) in conventional method vs ultrasound-guided method
The occurrence of dialysis incidents caused by catheters dysfunction | During procedure
  Compare the occurrence of dialysis incidents caused by catheters dysfunction (decrease in dialysis flow, single-puncture dialysis, shortening of dialysis time, loss of circuit) in conventional method vs ultrasound-guided method
Patient satisfaction | 30 days, 90 days, 180 days and 12 months after enrollment
  Compare the patient satisfaction in conventional method vs ultrasound-guided method using a satisfaction questionnaire
Patient comfort | During the procedure
  Compare the patient comfort in conventional method vs ultrasound-guided method. The visual analogue scale (VAS) will be used by patients > 5 years of age. The VAS measures from 0 to 10 the intensity of pain. The higher the score the less comfortable the procedure
Patient comfort | During the procedure
  Compare the patient comfort in conventional method vs ultrasound-guided method. The neonatal pain and discomfort scale (EDIN Échelle Douleur Inconfort Nouveau-Né ) will be used by patients ≤ 5 years of age.
  The EDIN scale uses five behavioural indicators of pain: facial activity, body movements, quality of sleep, quality of contact with nurses, and consolability.
  The scale measures friom 0 to 15 the intensity of pain. The higher the score the less comfortable the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jean Philippe BOUDET, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No